CLINICAL TRIAL: NCT05410613
Title: Effect of Combined Electromagnetic Field and a Plantar Resistance Exercise on Healing of Venous Leg Ulcer
Brief Title: Combined Electromagnetic Field and a Plantar Resistance Exercise With Venous Leg Ulcer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mona Mohamed Taha (Other)
Responsible Party: Sponsor-Investigator, Mona Mohamed Taha, associate professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P.T REC/012/003629
Record Dates: First submitted 2022-03-14; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer | interventions — Electromagnetic Fields

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- combined electromagnetic field and a plantar resistance (Experimental)
  Interventions: Combination Product: electromagnetic field and a plantar resistance exercise
- electromagnetic field (Experimental)
  Interventions: Device: Pulsed electromagnetic field
- conservative treatment for the ulcer (Active Comparator)
  Interventions: Other: usual care

INTERVENTIONS:
Combination Product: electromagnetic field and a plantar resistance exercise — Pulsed electromagnetic field therapy applied with intensity equal to 3mt and frequency of magnetic field impulses equal to 4 Hz.
  a plantar resistance exercise therapy by the StepIt rocker pedal, the overall exercise program will be to exercise on the pedal with the index leg for 1 min - then rest it for 1min - and to repeat this 10 times (20 minutes). This regime will be done twice daily (e.g .morning and evening).
  Arms: combined electromagnetic field and a plantar resistance
Device: Pulsed electromagnetic field — Pulsed electromagnetic field therapy applied with intensity equal to 3mt and frequency of magnetic field impulses equal to 4 Hz
  Arms: electromagnetic field
Other: usual care — standard general advice according to hospital protocol
  Arms: conservative treatment for the ulcer

SUMMARY:
The purpose of this study will investigate the effects of combined electromagnetic field and a plantar resistance exercise therapy versus electromagnetic field on healing of venous leg ulcer .

ELIGIBILITY:
Inclusion Criteria:

patients with venous leg ulcer

Exclusion Criteria:

patients who have one or more of the following conditions:

* peripheral vascular disease (PVD), (ABPI<0.8).
* venous leg ulcers with cellulitis or infection symptoms, as well as venous leg ulcers with necrotic tissue or slough or had more than one ulcer.
* other types of ulcers, such as rheumatoid vasculitis, diabetic foot, and malignant ulceration; corticosteroids use ; patients with dementia or who were disoriented;
* undertaken another physical therapy modality for ulcer healing.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-06-20 (Estimated)

PRIMARY OUTCOMES:
Ulcer surface area | two months
  Ulcer surface (UAS) would be calculated by placing a piece of sterilized transparency film over the ulcer and tracing the ulcer perimeter on the film with fine tipped transparency marker.
Ulcer volume measurement | two months
  Ulcer volume : The ulcer would be traced on transparent paper and placed over the metric graph paper to have the longest length and width.
  * A disposable measuring tape would be directed into the deepest point of the ulcer to record the ulcer depth.
  * (Width x length x depth) would be calculated to have the volume of the ulcer
Pressure Ulcer Scale for Healing (PUSH) | two months
  Categorize the ulcer with respect to surface area, exudate, and type of wound tissue

CONTACTS AND LOCATIONS:
Overall Officials: ASMAA FAWZY EL-SAYED, lecturer, Principal Investigator — Surgical department-Mansoura Health Insurance Hospital
Locations (1):
- Surgical department-Mansoura Health Insurance Hospital, Al Mansurah, Egypt